CLINICAL TRIAL: NCT04463056
Title: A Multicenter, Open Label, Randomized, Parallel-group Study of Efficacy and Safety of Eculizumab (JSC GENERIUM, Russia) vs. Soliris® (Alexion Pharma GmbH, Switzerland) in Patients With Paroxysmal Nocturnal Hemoglobinuria
Brief Title: Efficacy and Safety of Elizaria® vs. Soliris® in Patients With PNH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECU-PNH-III; #546 eff date 17.10.2017 (Other: Ministry of Health of Russia)
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2018-10

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; Marchiafava-Micheli Syndrome; Paroxysmal Hemoglobinuria
Keywords: Paroxysmal Cold Hemoglobinuria; eculizumab; Complement Inactivating Agents; Hemolysis; Anemia, Hemolytic; Anemia; Hematologic Diseases; Bone Marrow Diseases; Hemoglobinuria; Proteinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis; Anemia, Hemolytic; Anemia; Hematologic Diseases; Bone Marrow Diseases; Hemoglobinuria; Proteinuria | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elizaria® (Experimental): International nonproprietary name: eculizumab
  Interventions: Biological: Elizaria®
- Soliris® (Active Comparator): International nonproprietary name: eculizumab
  Interventions: Biological: Soliris®

INTERVENTIONS:
Biological: Elizaria® — Induction cycle: 600 mg (2 vials of 30 mL, 10 mg/mL) intravenous infusion for 30 minutes once a week for 4 weeks. Maintenance therapy: 900 mg (3 vials of 30 mL, 10 mg/mL) intravenous infusion for 30 minutes in Week 5, followed by 900 mg every 14 days.
  Other Names: eculizumab
  Arms: Elizaria®
Biological: Soliris® — Induction cycle: 600 mg (2 vials of 30 mL, 10 mg/mL) intravenous infusion for 30 minutes once a week for 4 weeks. Maintenance therapy: 900 mg (3 vials of 30 mL, 10 mg/mL) intravenous infusion for 30 minutes in Week 5, followed by 900 mg every 14 days.
  Other Names: eculizumab
  Arms: Soliris®

SUMMARY:
It is a multicenter, open-label, randomized, parallel-group study of the efficacy and safety of Elizaria® (eculizumab, GENERIUM JSC, Russia) versus Soliris® (Alexion Pharma GmbH, Switzerland) in patients with paroxysmal nocturnal hemoglobinuria.

DETAILED DESCRIPTION:
After screening, patients meeting all of the inclusion / non-inclusion criteria and vaccinated against meningococcal infections were divided into two subgroups according to the eculizumab treatment status (Soliris® naïve patients / patients who had received Soliris® at a maintenance dose prior to the trial inclusion). Each subgroup included an even number of patients to maintain recruitment balance. Then, patients of each subgroup were distributed into one of two treatment groups by the method of stratified block randomization at a 1:1 ratio into groups A and B, respectively. In the first group (Group A), patients received infusions of Elizaria (eculizumab, GENERIUM JSC), in the second one (Group B) - infusions of Soliris®.

The duration of participation of each patient in the study, including the screening period, was about 30 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for participation in the study.
2. Men and women aged 18 to 65 years at the time of signing the Informed Consent Form.
3. Established diagnosis of paroxysmal nocturnal hemoglobinuria (PNH), confirmed by flow cytometry assessing the PNH red blood cell and white blood cell clone size, with intravascular hemolysis and current or previous concomitant clinical symptoms, irrespective of the need for blood transfusions and without signs of other disorders associated with bone marrow failure.
4. For patients, who have not received Soliris® before inclusion in this study: lactate dehydrogenase (LDH) level 1.5 times the upper limit of normal or higher as assessed by the central laboratory.
5. The patients receiving anticoagulants must take them at a stable dose for at least 4 weeks prior to screening. Patients receiving warfarin must have a stable international normalized ratio (INR) value. To confirm INR value stability, the patients have to provide a blood INR test at least 4 weeks prior to screening. The second INR assessment will be performed at the screening visit.
6. Documented vaccination against meningococcal infections (Neisseria meningitidis serogroups A, C, Y and W-135) the protective immunity of which did not wear off, at least 14 days prior to the administration of the first dose of the test or reference drug and the patient's consent for revaccination against meningococcal infections (Neisseria meningitidis serogroups A, C, Y and W-135) during participation in the current study if the protection from previous vaccination wears off.
7. Subjects' consent to use reliable contraceptive methods (the combination of at least 2 methods, including barrier contraception, for example, condoms with spermicide) from signing the Informed Consent Form for up to 10 weeks after stopping therapy.

Exclusion Criteria:

1. Hypersensitivity to the test drug, reference drug and their components.
2. Hypersensitivity to the active substance or any other component of the vaccine used to prevent meningococcal infection or a lifethreatening reaction to a previously administered vaccine containing similar ingredients.
3. Conditions associated with bone marrow failure and PNH clone (aplastic anemia, myelodysplastic syndrome, idiopathic myelofibrosis).
4. A history of infections caused by Neisseria meningitides.
5. Active systemic bacterial, viral, or fungal infection within 14 days prior to the administration of the first dose of the test or reference drug.
6. Fever of 38°С or higher within 7 days prior to the administration of the first dose of the test or reference drug.
7. Hereditary complement deficiencies.
8. Patients planning to undergo or with a history of bone marrow transplantation.
9. Initial treatment cycle (induction phase) of Soliris®; completed treatment with Soliris® less than 70 days before study inclusion, not related to the current study participation.
10. Vaccination with any live vaccine within 1 month prior to the administration of the first dose of the test or reference drug;
11. Concomitant diseases and conditions which may, in the Investigator's opinion, compromise the patient's safety in case of participation in the study or which could affect the safety data analysis in case of an exacerbation of this disease/condition during the study, including the following:

    * Myocardial infarction or stroke within the last 3 months, severe arrhythmia, NYHA functional class III/IV heart failure;
    * Psychiatric disorders;
    * Immune and endocrine disorders which are not controlled with medications (including decompensated diabetes mellitus and thyroid disorders);
    * Hematologic disorders requiring chemotherapy;
    * Current or prior oncologic disorders, except for successfully treated basal cell carcinoma;
    * Decompensated liver diseases.
12. Acquired immunodeficiency syndrome or human immunodeficiency virus (HIV) infection confirmed by test results.
13. Active viral hepatitis B and/or C at screening with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels 5 times the upper limit of normal or higher.
14. Positive syphilis test results.
15. Body mass index (BMI) ≤17 kg/m2 or ≥30 kg/m2.
16. Pregnancy or breastfeeding.
17. History of tuberculosis, alcohol addiction, medication abuse, or drug addiction.
18. Patient's participation in any clinical studies and/or using of not approved medications in the Russian federation within 30 days before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Area under the LDH concentration-time curve (LDH AUC) during the maintenance therapy with the test drug or the reference drug | week 22

SECONDARY OUTCOMES:
Area under the LDH concentration-time curve (LDH AUC) during 26-week therapy with the test product or the reference product | week 26
Hemoglobin level change during the maintenance therapy with the test drug or the reference drug | week 22
Number/proportion of the patients with stable hemoglobin level during the maintenance therapy with the test drug or the reference drug | week 22
Number/proportion of patients with various thrombotic complications developing during treatment with the test product or the reference product. | week 26
Number/proportion of patients who needed donor red blood cell transfusions during treatment with the test product or the reference product. | week 26
Number of donor red blood cell transfusions during treatment with the test product or the reference product. | week 26
Number/proportion of patients with breakthrough hemolysis | week 26
  Breakthrough hemolysis defined as at least one new episode or worsening of at least one previous signs of intravascular hemolysis (fatigue, hemoglobinuria, abdominal pain, dyspnea, severe vascular complications (including thrombosis), dysphagia or erectile dysfunction) associated with increased LDH after a previous decrease during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — AO GENERIUM
Locations (4):
- Russia (4):
  - Federal State Budget Funded Institution National Medical Research Center of Hematology, Ministry of Health of the Russian Federation (MoH of Russia), Moscow
  - Moscow State Budget Funded Healthcare Institution S. P. Botkin City Clinical Hospital, Moscow Department of Healthcare, Moscow
  - State Budget Funded Institution of Higher Education Academician I. P. Pavlov Saint-Petersburg State Medical University of the Ministry of Health of the Russian Federation, Saint Petersburg
  - State Budgetary Educational Institution of Higher Professional Education Samara State Medical University, Ministry of Health of the Russian Federation., Samara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kulagin AD, Ptushkin VV, Lukina EA, Davydkin IL, Korobkin AV, Shamrai VS, Konstantinova TS, Kaporskaya TS, Mitina TA, Ksenzova TI, Zuev EV, Markova OA, Gapchenko EV, Kudlay DA. Randomized multicenter noninferiority phase III clinical trial of the first biosimilar of eculizumab. Ann Hematol. 2021 Nov;100(11):2689-2698. doi: 10.1007/s00277-021-04624-7. Epub 2021 Aug 16. PMID 34398258
- See also: Kulagin, A.D., Ptushkin, V.V., Lukina, E.A. et al. Randomized multicenter noninferiority phase III clinical trial of the first biosimilar of eculizumab. Ann Hematol (2021). https://doi.org/10.1007/s00277-021-04624-7 — https://link.springer.com/article/10.1007/s00277-021-04624-7#citeas